CLINICAL TRIAL: NCT03069885
Title: Incisional Negative Pressure Wound Therapy (Prevena™) vs. Conventional Post-operative Dressing After Immediate Breast Reconstruction; a Randomized Controlled Clinical Trial
Brief Title: iNPWT in Immediate Breast Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 52373
Record Dates: First submitted 2017-02-20; First posted 2017-03-03 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Breast Neoplasm Female; Mammaplasty

STUDY DESIGN:
Intervention Model Description: The project is conducted as a randomized controlled trial. Patients included in the study will be randomized to either conventional post-operative dressing or PrevenaTM iNPWT treatment. Patients are allocated in a 1:1 ratio, with 30 patients treated with PrevenaTM and 30 patients treated with conventional post-operative dressing.
Masking Description: The study will not be blinded, since the PrevenaTM-device makes a sound, when generating negative pressure, and the dressing looks a lot different compared to the conventional post-operative dressing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard postoperative dressing group (Active Comparator): 30 patients treated with conventional post-operative dressing.
  Interventions: Other: Standard Postoperative dressing
- Prevena group (Experimental): 30 patients treated with PrevenaTM (incisional negative pressure wound therapy)
  Interventions: Device: Prevena

INTERVENTIONS:
Device: Prevena — Incisional negative pressure wound therapy (iNPWT), is a new approach for surgical site closure using negative pressure wound therapy (NPWT). Recently, PrevenaTM have been approved as an iNPWT-system applied at the end of surgery, while still in a sterile environment. PrevenaTM consist of a sponge foam with a bactericidal silver lining dressed with an adherent film, connected to a vacuum device, producing a vacuum of 125 mm Hg. The PrevenaTM foam and dressing is placed over the suture line, and is recommended to be kept in place for a continuous period lasting between 2 and 7 days.
  Arms: Prevena group
Other: Standard Postoperative dressing — The standard postoperative dressing, using steri strips placed over the suture line.
  Arms: Standard postoperative dressing group

SUMMARY:
Due to the Danish breast cancer-screening programme and the increased use of genetic counselling, Danish women are being diagnosed with breast cancer, or a high lifetime risk of developing breast cancer, at a younger age than previously. An increasing proportion of these women pursue an immediate breast reconstruction, where the breast is removed and reconstructed in a single surgical procedure.

As some of these women will need to undergo adjuvant cancer therapy after their breast surgery, fast recovery is essential in order for the adjuvant therapy not to be delayed. With the development of new surgical techniques, the complication rate to the immediate breast reconstructions has improved. However, wound-healing issues remain one of the most common complications to the surgery with the possibility of delaying the adjuvant therapy and diminish the aesthetic result.

Incisional negative pressure wound therapy (iNPWT), is a new approach for surgical site closure. Recently, iNPWT has shown promising results in lowering post-operative complications, including wound-healing issues, in other surgical settings. However, iNPWT has still not been studied in an immediate breast reconstructive setting.

The current randomized controlled clinical study will investigate if an iNPWT system, is able to provide women seeking an immediate breast reconstruction with faster healing and superior aesthetic results compared to the conventional post-operative wound dressings used today. The investigators plan to include 60 women, randomized in a 1:1 ratio between iNPWT or conventional wound dressing. The primary outcome measure is the time until removal of the surgical drains, which corresponds to the healing progression. Secondarily, complications to the surgery, assessment of the scar (measured using the Patient and Observer Scar Assessment Scale) and patient reported satisfaction with the reconstruction (assessed using the BREAST-Q questionnaire) will be performed. Included patients are examined pre-operatively, and at the routine controls at four weeks and four months post operatively.

The results from the current study will elucidate if iNPWT aids wound healing after immediate breast reconstruction, which would lead to fewer patients experiencing delays before their adjuvant therapy. Furthermore, the results from the aesthetic satisfaction will elucidate if iNPWT provides the patients with a better self-reported aesthetic result.

DETAILED DESCRIPTION:
Incisional negative pressure wound therapy (Prevena™) vs. conventional post-operative dressing after immediate breast reconstruction; a randomized controlled clinical trial.

• Introduction

Over the last 60 years, there has been a steady rise in the incidence of breast cancer in Denmark. Due to the Danish breast cancer screening program and the increasing use of genetic counseling, patients are diagnosed with breast cancer, pre-cursors hereof, or an increased lifetime risk of breast cancer at an earlier age than previously. In women with high estimated risk of breast cancer, current studies indicate a reduced lifetime risk of cancer, and thereby increased survival, when undergoing a risk reducing mastectomy. Therefore, Danish women may choose to undergo a risk reducing mastectomy, if they have a estimated lifetime risk of breast cancer at 30% or above.

At the Department of Plastic and Breast Surgery, Aarhus University Hospital, Denmark, there has been a rise in the number of immediate breast reconstructions performed, currently counting approximately 200 per year. This increase is partly due to the increasing number of prophylactic risk reducing mastectomies, as well as an increasing number of women choosing immediate breast reconstruction when diagnosed with Ductal Carcinoma In-Situ (DCIS).

As some of these women will need to undergo adjuvant cancer therapy after their breast surgery, fast recovery is essential in order for the adjuvant therapy to not be delayed.

Women undergoing surgery at a younger age, will presumably live for a longer time, with possible complications of the immediate breast reconstruction. Therefore, a good result at the first surgery and fast rehabilitation, are of essential importance for these women's recovery and quality of life.

The immediate breast reconstruction, holds several benefits compared to mastectomy and subsequent delayed breast reconstruction. Benefits such as rapid return to work, low complication rate, good aesthetic outcome, and the need for only one surgery, but the surgery is not free of complications. The complication rate in immediate breast reconstruction, is reported in the range of 3,9% to 14,8 %, with the most frequent complications being skin necrosis, surgical site infections (SSI), implant loss and haematoma/seroma.

Incisional negative pressure wound therapy (iNPWT), is a new approach for surgical site closure using negative pressure wound therapy (NPWT). Recently, PrevenaTM have been approved as an iNPWT-system applied at the end of surgery, while still in a sterile environment. PrevenaTM consist of a sponge foam with a bactericidal silver lining, dressed with an adherent film, connected to a vacuum device, producing a vacuum of 125 mm Hg. The PrevenaTM foam and dressing is placed over the suture line, and is recommended to be kept in place for a continuous period lasting between 2 and 7 days.

iNPWT is based on the principles behind NPWT, most known as vacuum assisted closure (V.A.C.), which is well described in the literature.

NPWT has been shown to be an efficient way of treating chronic wounds, by increasing blood flow and formation of granulation tissue, stimulate cell proliferation and angiogenesis, decrease bacterial count, reduce oedema, improve wound closure rates, collagen organization and wound maturation in animal- and clinical-studies.

Furthermore, recently iNPWT has shown promising results in lowering post-operative complications, with lower rate of surgical site infection, lower incidence of wound dehiscence, and lower loss of split thickness skin grafts.

In an experimental porcine setup, indications of increased lymph clearance with lower production of seroma/hematoma has been shown when using iNPWT. Additionally, in a biomechanical analysis, Wilkes et al. found evidence of reduced lateral stress on wounds, which in theory, could lead to faster closure and improved scar aesthetics.

Overall, iNPWT has been shown to reduce several of the most frequent complications that may occur following an immediate breast reconstruction. However, in an immediate breast reconstructive setting, iNPWT has not yet been studied, and in breast surgery in general, there is only limited data on the use of NPWT and iNPWT.

The current study aims to investigate whether PrevenaTM provides a superior post-operative wound treatment, when compared to conventional treatment, for women undergoing a prophylactic or therapeutic mastectomy with an immediate breast reconstruction.

• Hypothesis

iNPWT, administrated by PrevenaTM, will reduce the post-operative complications in patients undergoing immediate breast reconstruction, compared to conventional post-operative dressing.

• Aim

The aim of the current study is to evaluate whether iNPWT provides superior wound treatment for patients undergoing an immediate breast reconstruction, compared to treatment with conventional post-operative dressing. The results from this study will possibly help to minimize the complication rate and increase the patient satisfaction, by finding the optimal wound treatment for immediate breast reconstructions and thereby contributing to a faster recovery, for women who undergo this procedure.

• Methods

The project is conducted as a randomized controlled trial. Patients included in the study will be randomized to either conventional post-operative dressing or PrevenaTM iNPWT treatment. Patients are allocated in a 1:1 ratio, with 30 patients treated with PrevenaTM and 30 patients treated with conventional post-operative dressing.

* Study population

  60 patients admitted for immediate breast reconstruction at the Department of Plastic Surgery, Aarhus University Hospital, will upon informed consent be offered participation in this prospective, randomized study using two types of post-operation dressing after the breast reconstruction surgery
* Risks, side effects and disadvantages

As with all surgery, there is a risk of wound infection, blood clots and altered sensation in the operated area. This can lead to antibiotic treatment, or where appropriate, a second surgery to stop bleeding or remove damaged tissue. These risks are, however, associated with the breast reconstruction itself, and not associated with participating in the research project.

PrevenaTM have been approved and used internationally as a post-operative dressing since 2010. PrevenaTM is well described in the medical literature, achieving good results compared to conventional post-operative dressing, showing fewer, or the same amount of complications. The risks for the patients choosing to participate in the project are thus solely related to the breast reconstruction itself, and not to the participation in the research project.

• Economics

Initiators of this project are the Department of Plastic and Brest Surgery, Aarhus University Hospital. All costs of the investigated post-surgical wound treatment (PrevenaTM or conventional post-operative treatment) are held by the Department of Plastic and Brest Surgery, Aarhus University Hospital. Participating patients are not given any reimbursement. Patients may, however, apply for reimbursement to cover documented travel expenses, in regards to the regulations of the Central Denmark Region.

The salary for the scientific personnel, and cost of materials and conferences will be sought covered by external funding from private and/or governmental funds. Funding will solely be sought from foundations and scholarships, where the benefactors do not have a financial interest in the outcome of the study. Furthermore, funding will only be sought from sources, where the research project can remain independent from the contributor.

• Publication

Positive, negative, as well as inconclusive results are expected to be published in a peer-reviewed international journal with interest in the field. Furthermore, the results are expected to be presented at a national or international conference in plastic and reconstructive surgery.

• Ethical considerations

It is expected that the number of women seeking an immediate breast reconstruction will increase. The proposed study will aid in finding the most optimal wound dressing following this surgery. Conducting studies that help bring down the complication rates for these types of surgery is of utmost importance, both for the individual patient undergoing the surgery and in a socio-economic setting.

All of the patients invited to participate in this study has been evaluated by experienced breast and plastic surgeons to be best suited with an immediate breast reconstruction with implant.

PrevenaTM, or iNPWT, have shown good results in previous studies in other types of surgery, showing none or only minor complications. The general treatment, using steri strips, has been used for many years as the primary choice.

As the investigators expect fewer or the same amount of complications when using PrevenaTM, there is no predictable disadvantage for the individual patient in regards to participating in the study.

The patients' privacy, physical and mental integrity and the Danish law concerning the processing of personal data will be respected. Furthermore, the research project will be carried out in accordance with the Helsinki Declaration II.

The project is approved by the Central Denmark Regional Committee on Health Research Ethics, see appendix 2 (in Danish) and registered at the Central Denmark Regions joint application for the Danish Data Protection Agency, see Appendix 3 (in Danish).

• Perspectives

The results from the current study will elucidate if iNPWT aids wound healing after immediate breast reconstruction, which would lead to fewer patients experiencing delays before their adjuvant therapy. Furthermore, the results from the aesthetic satisfaction will elucidate if iNPWT provides the patients with a better self-reported aesthetic result.

Faster healing could potentially result in a shorter hospital stay. At the Department of Plastic and Breast Surgery, Aarhus University Hospital, the approximate cost per hospitalization day is 4000 Danish kroner (DKK). With a price of 975 DKK., the PrevenaTM-device could be a potential economical benefit, with an average reduction in hospitalization time by just a single day. Finally, the potential cost savings do to fewer post-operative complications, should be held in consideration.

All in all, the results from the current study may provide the increasing number of women undergoing an immediate breast reconstruction with a shorter hospital stay, a better breast reconstructive result and faster adjuvant therapy.

ELIGIBILITY:
60 patients admitted for immediate breast reconstruction at the Department of Plastic Surgery, Aarhus University Hospital, will upon informed consent be offered participation in this prospective, randomized study using two types of post-operation dressing after the breast reconstruction surgery.

Inclusion Criteria:

* Patient deemed best suited with an immediate breast reconstruction using implant by the consultant plastic- and breast surgeon.
* Patient is older than 18 years of age.
* Patient understand enough Danish to comprehend the given information and to complete the study questionnaires.

Exclusion Criteria:

* Current smokers (patients not having paused for a minimum of four weeks prior to surgery)
* Non-eligible patients, as assessed by the operating surgeon
* High level of co-morbidity, as assessed by operating surgeon or anaesthesiologist
* Allergic to band-aids.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Drain time | 1-14 days after surgery
  Time to removal of surgical drains.

SECONDARY OUTCOMES:
Surgical site infection | 1-30 days after surgery
  Post-operative surgical site infection rate
Skin necrosis | 1-30 days after surgery
  Rate of skin necrosis in relation to the breast reconstruction
Hospitalization time | 1-30 days after surgery
  Post-operation hospitalization time
Patient and observer assessment of the scars | 4 weeks and 4 month after surgery
  The quality and appearance of the scar will be investigated at the post-operative clinical control by using the Patient and observer Scar Assessment Scale (POSAS). The POSAS is an instrument designed to measure scar quality. It consists of two scales, one completed by the patient and one completed by the observer
Patient satisfaction and quality of Life | 1 week before surgery until 4 months after surgery
  Patients included in the study will be asked to complete the BREAST-Q pre-reconstruction module before their breast reconstruction, and the BREAST-Q post-reconstruction module at the post-operative clinical control. The BREAST-Q is a patient reported outcome measure tool specifically designed and validated for use in breast reconstruction patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tine E Damsgaard, MD, Phd., Study Director — University of Aarhus and Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, NBG, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meijers-Heijboer H, van Geel B, van Putten WL, Henzen-Logmans SC, Seynaeve C, Menke-Pluymers MB, Bartels CC, Verhoog LC, van den Ouweland AM, Niermeijer MF, Brekelmans CT, Klijn JG. Breast cancer after prophylactic bilateral mastectomy in women with a BRCA1 or BRCA2 mutation. N Engl J Med. 2001 Jul 19;345(3):159-64. doi: 10.1056/NEJM200107193450301. PMID 11463009
- [Background] Skytte AB, Cruger D, Gerster M, Laenkholm AV, Lang C, Brondum-Nielsen K, Andersen MK, Sunde L, Kolvraa S, Gerdes AM. Breast cancer after bilateral risk-reducing mastectomy. Clin Genet. 2011 May;79(5):431-7. doi: 10.1111/j.1399-0004.2010.01604.x. Epub 2011 Jan 4. PMID 21199491
- [Background] Colwell AS, Damjanovic B, Zahedi B, Medford-Davis L, Hertl C, Austen WG Jr. Retrospective review of 331 consecutive immediate single-stage implant reconstructions with acellular dermal matrix: indications, complications, trends, and costs. Plast Reconstr Surg. 2011 Dec;128(6):1170-1178. doi: 10.1097/PRS.0b013e318230c2f6. PMID 22094736
- [Background] Salzberg CA, Ashikari AY, Koch RM, Chabner-Thompson E. An 8-year experience of direct-to-implant immediate breast reconstruction using human acellular dermal matrix (AlloDerm). Plast Reconstr Surg. 2011 Feb;127(2):514-524. doi: 10.1097/PRS.0b013e318200a961. PMID 21285756
- [Background] Bollero D, Malvasio V, Catalano F, Stella M. Negative pressure surgical management after pathological scar surgical excision: a first report. Int Wound J. 2015 Feb;12(1):17-21. doi: 10.1111/iwj.12040. Epub 2013 Feb 19. PMID 23418720
- [Background] Morykwas MJ, Argenta LC, Shelton-Brown EI, McGuirt W. Vacuum-assisted closure: a new method for wound control and treatment: animal studies and basic foundation. Ann Plast Surg. 1997 Jun;38(6):553-62. doi: 10.1097/00000637-199706000-00001. PMID 9188970
- [Background] Jacobs S, Simhaee DA, Marsano A, Fomovsky GM, Niedt G, Wu JK. Efficacy and mechanisms of vacuum-assisted closure (VAC) therapy in promoting wound healing: a rodent model. J Plast Reconstr Aesthet Surg. 2009 Oct;62(10):1331-8. doi: 10.1016/j.bjps.2008.03.024. Epub 2008 Jul 9. PMID 18617451
- [Background] Argenta LC, Morykwas MJ. Vacuum-assisted closure: a new method for wound control and treatment: clinical experience. Ann Plast Surg. 1997 Jun;38(6):563-76; discussion 577. PMID 9188971
- [Background] Saxena V, Hwang CW, Huang S, Eichbaum Q, Ingber D, Orgill DP. Vacuum-assisted closure: microdeformations of wounds and cell proliferation. Plast Reconstr Surg. 2004 Oct;114(5):1086-96; discussion 1097-8. doi: 10.1097/01.prs.0000135330.51408.97. PMID 15457017
- [Background] Greene AK, Puder M, Roy R, Arsenault D, Kwei S, Moses MA, Orgill DP. Microdeformational wound therapy: effects on angiogenesis and matrix metalloproteinases in chronic wounds of 3 debilitated patients. Ann Plast Surg. 2006 Apr;56(4):418-22. doi: 10.1097/01.sap.0000202831.43294.02. PMID 16557076
- [Background] Gomoll AH, Lin A, Harris MB. Incisional vacuum-assisted closure therapy. J Orthop Trauma. 2006 Nov-Dec;20(10):705-9. doi: 10.1097/01.bot.0000211159.98239.d2. PMID 17106382
- [Background] Stannard JP, Volgas DA, McGwin G 3rd, Stewart RL, Obremskey W, Moore T, Anglen JO. Incisional negative pressure wound therapy after high-risk lower extremity fractures. J Orthop Trauma. 2012 Jan;26(1):37-42. doi: 10.1097/BOT.0b013e318216b1e5. PMID 21804414
- [Background] Chadi SA, Kidane B, Britto K, Brackstone M, Ott MC. Incisional negative pressure wound therapy decreases the frequency of postoperative perineal surgical site infections: a cohort study. Dis Colon Rectum. 2014 Aug;57(8):999-1006. doi: 10.1097/DCR.0000000000000161. PMID 25003295
- [Background] Llanos S, Danilla S, Barraza C, Armijo E, Pineros JL, Quintas M, Searle S, Calderon W. Effectiveness of negative pressure closure in the integration of split thickness skin grafts: a randomized, double-masked, controlled trial. Ann Surg. 2006 Nov;244(5):700-5. doi: 10.1097/01.sla.0000217745.56657.e5. PMID 17060762
- [Background] Kilpadi DV, Cunningham MR. Evaluation of closed incision management with negative pressure wound therapy (CIM): hematoma/seroma and involvement of the lymphatic system. Wound Repair Regen. 2011 Sep-Oct;19(5):588-96. doi: 10.1111/j.1524-475X.2011.00714.x. PMID 22092797
- [Background] Wilkes RP, Kilpad DV, Zhao Y, Kazala R, McNulty A. Closed incision management with negative pressure wound therapy (CIM): biomechanics. Surg Innov. 2012 Mar;19(1):67-75. doi: 10.1177/1553350611414920. Epub 2011 Aug 25. PMID 21868417
- [Background] Kostaras EK, Tansarli GS, Falagas ME. Use of negative-pressure wound therapy in breast tissues: evaluation of the literature. Surg Infect (Larchmt). 2014 Dec;15(6):679-85. doi: 10.1089/sur.2013.165. PMID 24871230
- [Background] Doig GS, Simpson F. Randomization and allocation concealment: a practical guide for researchers. J Crit Care. 2005 Jun;20(2):187-91; discussion 191-3. doi: 10.1016/j.jcrc.2005.04.005. PMID 16139163
- [Background] Pusic AL, Klassen AF, Scott AM, Klok JA, Cordeiro PG, Cano SJ. Development of a new patient-reported outcome measure for breast surgery: the BREAST-Q. Plast Reconstr Surg. 2009 Aug;124(2):345-353. doi: 10.1097/PRS.0b013e3181aee807. PMID 19644246
- [Background] van de Kar AL, Corion LU, Smeulders MJ, Draaijers LJ, van der Horst CM, van Zuijlen PP. Reliable and feasible evaluation of linear scars by the Patient and Observer Scar Assessment Scale. Plast Reconstr Surg. 2005 Aug;116(2):514-22. doi: 10.1097/01.prs.0000172982.43599.d6. PMID 16079683
- [Background] Kim SY, Lim SY, Mun GH, Bang SI, Oh KS, Pyon JK. Evaluating the effectiveness of cryopreserved acellular dermal matrix in immediate expander-based breast reconstruction: a comparison study. Arch Plast Surg. 2015 May;42(3):316-20. doi: 10.5999/aps.2015.42.3.316. Epub 2015 May 14. PMID 26015887
- See also: NORDCAN (Association of the Nordic Cancer Registries). Cancer stat fact sheets Denmark - Breast. 2015. — http://www-dep.iarc.fr/NORDCAN/DK/StatsFact.asp?cancer=200&country=208
- See also: DBCG (Danish Breast Cancer Cooperative Group)-retningslinier 2010 - Kapitel 19: Genetisk udredning, rådgivning og molekylærgenetisk analyse. 2010. — http://www.dbcg.dk/PDF%20Filer/Retningslinier%202010%20Kap%2019%20010410.pdf